CLINICAL TRIAL: NCT04311853
Title: Pilot Study of Type 2 Diabetes Evidence-Based Nutrition Practice Guidelines--Field Test of Toolkit and Preliminary Outcomes
Brief Title: Evidence-Based Nutrition Practice Guidelines of Toolkit and Preliminary Outcomes
Status: Completed | Type: Observational
Sponsor: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Alison L Steiber, Chief Science Officier, Academy of Nutrition and Dietetics
Other Study IDs: not determined yet
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- practitioner interviews: phone interviews conducted

SUMMARY:
The goal of this study is to field test ADA's Type 2 Diabetes Evidence-Based nutrition Practice Guidelines (EBNPG) for Adults in 2008 as a tool for registered dietitians (RDs) for their patients with with type 2 diabetes who have no evidence of organ damage. A six month pilot study will be conducted to determine the feasibility of training RDs in documenting the outcomes of implementing Medical Nutrition Therapy (MNT) using ADA's evidence-based GL for T2D.

ELIGIBILITY:
Inclusion Criteria:

* over 19 years
* no documented claims for the treatment of TD over the past 7 years
* no MNT claims submitted within the past 12 months
* not under RD care
* able to make visits to the clinic per guidelines

Exclusion Criteria:

* not in end-stage renal disease or renal insufficiency; history of Cardiovascular Disease,Chronic Athrosclerotic Disease, or Myocardial Infection; Chronic Obstructive Pulmonary Disease, untreated depression, severe psychiatric illness; cancer diagnosis in previous two years or on-going radiation or chemotherapy treatment; Congestive Heart Failure.
* pregnant or lactating at time of study
* presence of cognitive limitations that preclude making lifestyle or dietary changes as assessed by the RD during the initial interview

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: practitioners working with patients who have heart failure
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Implementation of new evidence-based nutrition practice guidelines | six months
  RDs and RDs with CDE credential, will have reached the target professional goals in successful implementation of new evidence-based nutrition practice guidelines in daily clinical practice.

SECONDARY OUTCOMES:
Improved health outcomes | six months
  Patients counseled by either an RD, or an RD with CDE credential, will exhibit improvements in critical health outcomes, relative to baseline levels.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Snetselaar, PhD, RD, LD, Principal Investigator — University of Iowa; Esther F Myers, PhD, RD, Principal Investigator — Academy of Nutrition and Dietetics